CLINICAL TRIAL: NCT00724555
Title: Acute Stroke Program of Interventions Addressing Racial and Ethnic Disparities
Acronym: ASPIRE
Status: Completed | Type: Observational
Sponsor: Georgetown University (Other)
Collaborators: Medstar Health Research Institute (Other); Howard University (Other); George Washington University (Other); University of Michigan (Other); University of Wisconsin, Madison (Other); Johns Hopkins University (Other); University of Alabama at Birmingham (Other); MedStar Good Samaritan Hospital (Unknown); Union Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chelsea Kidwell, M.D., Professor of Neurology and Medical Director, Georgetown University Stroke Center, Georgetown University
Other Study IDs: U54NS057405_ASPIRE; 2007-439; U54NS057405 (NIH)
Record Dates: First submitted 2008-07-28; First posted 2008-07-29 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2014-01

CONDITIONS: Stroke
Keywords: stroke; tissue plasminogen activator; tPA
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Adults living in DC neighborhoods with high proportions of underserved adults. The age of the cohort members will reflect the age of DC residents who suffer most from stroke.

SUMMARY:
The purpose of this study is to increase treatment of acute stroke with tissue plasminogen activator (tPA) across the District of Columbia. This study, however, will not evaluate tPA as an intervention.

DETAILED DESCRIPTION:
There are a number of well-known barriers to receiving tissue plasminogen activator (tPA) including transit time to hospital, paramedic and provider training, tPA standing orders, and provider guidelines. Among underserved populations, limited stroke knowledge, socioculturally determined attitudes, and beliefs and myths held by community members may serve as additional barriers that hinder these populations from receiving tPA and acute stroke care. Targeted multilevel interventions designed to overcome specific barriers may significantly increase the number of individuals with stroke who are appropriately treated with intravenous tPA (IV tPA) in underserved communities. Identification of the specific components of healthcare interventions that are the most effective is critical to improve delivery of acute stroke therapy.

The goal of this study is to learn more about public knowledge, attitudes, beliefs and perceptions regarding stroke and stroke treatment in order to identify sociocultural and environmental barriers to receiving tPA and acute stroke care in an underserved community. This study will also determine if implementation of a multilevel intervention program can significantly increase the number of people with ischemic stroke who are appropriately treated with IV tPA in a predominantly underserved community.

In the study, researchers will evaluate the different levels of the intervention to determine which efforts are most effective.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of acute ischemic stroke
* over the age of 18

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult residents of the District of Columbia
Sampling Method: Non-Probability Sample
Enrollment: 2005 (Estimated)
Dates: Start 2008-02; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
The proportion of people with ischemic stroke appropriately treated with IV tPA. | 4 years

SECONDARY OUTCOMES:
Qualitative data collected from the community will identify baseline levels of knowledge, attitudes, and perceived and encountered barriers to acute stroke treatment. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Chelsea Kidwell, MD, Principal Investigator — Georgetown University
Locations (8):
- United States (8):
  - Georgetown University, ASPIRE Coordinating Center, Washington D.C., District of Columbia
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Providence Hospital, Washington D.C., District of Columbia
  - United Medical Center (formerly known as Greater Southeast Community Hospital), Washington D.C., District of Columbia
  - George Washington University Hospital, Washington D.C., District of Columbia
  - Howard University Hospital, Washington D.C., District of Columbia
  - Columbia University Medical Center, New York, New York

REFERENCES:
- [Derived] Boden-Albala B, Edwards DF, St Clair S, Wing JJ, Fernandez S, Gibbons MC, Hsia AW, Morgenstern LB, Kidwell CS. Methodology for a community-based stroke preparedness intervention: the Acute Stroke Program of Interventions Addressing Racial and Ethnic Disparities Study. Stroke. 2014 Jul;45(7):2047-52. doi: 10.1161/STROKEAHA.113.003502. Epub 2014 May 15. PMID 24876243